CLINICAL TRIAL: NCT04405752
Title: Evaluation of a New Metal Biliary Stent of 12-mm Diameter: a Case Control Study
Acronym: BIGDIAM
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: BIGDIAM-IPC 2018-056
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Malignant Biliary Obstruction
Keywords: biliary stent; malignant biliary stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 12-mm diameter metallic billiary stent
  Interventions: Device: 12-mm metallic biliary stent
- 10-mm diameter metallic billiary stent
  Interventions: Device: 10-mm metallic biliary stent

INTERVENTIONS:
Device: 12-mm metallic biliary stent — Metallic biliary stent, covered or uncovered,KEBOMED HILZO 12mm in diameter (length 4 or 6 cm).
  Groups: 12-mm diameter metallic billiary stent
Device: 10-mm metallic biliary stent — Biliary, metallic, covered or uncovered stent, COOK EVOLUTION 10mm in diameter (length 4 or 6 cm)
  Groups: 10-mm diameter metallic billiary stent

SUMMARY:
Biliary stent allows the drainage of the bile ducts palliatively or preoperatively in the event of malignant biliary stenosis, and a biliary calibration in the event of benign stenosis. Currently, by expert agreement, the diameter is 10-mm for metal stent. Since 2017, larger stents have been marketed in France and are approved for the biliary drainage of benign and malignant biliary stricture. These new 12-mm diameter stent could reduce the risk of recurrent biliary obstruction (RBO) and therefore increase the stent duration. The aim of our study was to compare whether the permeability of 12-mm diameter stent was better than a conventional 10-mm, covered or uncovered prosthesis depending on the indication.

ELIGIBILITY:
Inclusion Criteria:

* benign and malignant biliary stricture of the lower or median portion of the main biliary duct with indication of biliary stent placement including pre-operatively drainage
* age≥ 18 years old;
* Karnofsky score ≥ 40.

Exclusion Criteria:

* hilar stenosis;
* coagulation disorder (PT <50%, platelets < 80,000).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From April 2017 to April 2018, at the Paoli Calmettes Institute, 24 patients with benign or malignant biliary strictures were treated by placing a metallic biliary stent, covered or uncovered, KEBOMED HILZO 12mm in diameter (length 4 or 6 cm).
  "Control" patients, who had benefited from the placement of a biliary, metallic, covered or uncovered stent, COOK EVOLUTION 10mm in diameter (length 4 or 6 cm) were searched on a database (ConsortConsore®️)extending from January 2016 to March 2018. "Cases" patients were exactly matched in a ratio 1:2 to "control" on the following criteria: age (per decade), sex, pathology responsible for biliary stenosis (i.e., benign or malignant stenosis) and type of stent (i.e., covered/uncovered). When we searched for control patients in our database, the first patient with matching criteria was included.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Time to recurrent biliary obstruction (RBO) | 12 months
  RBO is defined as the time from the prosthesis deployment to until the first biliary stent obstruction (patency

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Caillol, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhône, France

IPD SHARING:
Plan to Share IPD: No